CLINICAL TRIAL: NCT05572073
Title: A Natural History Study in Individuals With Otoferlin Gene-mediated Hearing Loss
Brief Title: Otoferlin Gene-mediated Hearing Loss Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Akouos, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: AK-OTOF-NHS-002
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: Otoferlin Gene, sensorineural hearing loss (SNHL), auditory neuropathy, auditory neuropathy spectrum disorder
MeSH Terms: conditions — Hearing Loss, Sensorineural; Auditory neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective
  Interventions: Other: Natural History Study
- Prospective
  Interventions: Other: Natural History Study

INTERVENTIONS:
Other: Natural History Study — Natural History Study

SUMMARY:
This is a retrospective and prospective longitudinal study in participants with Otoferlin Gene-Mediated Hearing Loss.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical presentation of bilateral sensorineural hearing loss (SNHL), including auditory neuropathy (AN) / auditory neuropathy spectrum disorder (ANSD) phenotype or medical history of AN / ANSD phenotype earlier in life
2. Mutation(s) in the otoferlin gene
3. Able and willing to comply with all study requirements, as evidenced by successful completion of the informed consent (and assent, if applicable) process

   Additional Criteria for Inclusion in the Prospective Phase:
4. Presence of OAE / CM and absent / abnormal ABRs in at least one ear (that does not have a cochlear implant) within 12 months prior to or at the Month 0 visit

Exclusion Criteria:

1. Unwillingness or inability of the potential participant and/or legally authorized representative to comply with all protocol requirements
2. Presence of cochlear nerve deficiency and/or cochlear nerve dysplasia

   Additional Criteria for Exclusion from the Prospective Phase:
3. Presence of bilateral cochlear implants at the time of record review or planned within the next 6 months
4. Presence of middle ear or auditory brainstem implant(s) at the time of record review or planned within the next 6 months
5. Any condition that would not allow the potential participant to complete follow-up assessments during the course of the study and/or, in the opinion of the Investigator, makes the potential participant unsuitable for the study

Note: Potential participants will not be excluded based on their sex, gender, race, or ethnicity

Max Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with hearing loss due to confirmed otoferlin gene mutation(s)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
ABR | First audiologic data in participant medical record through five-year prospective follow up
  Auditory Brainstem Response

SECONDARY OUTCOMES:
OAE | First audiologic data in participant medical record through the five-year prospective follow up
  Otoacoustic Emissions

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Reape, MD, Study Director — Akouos, Inc.
Locations (10):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- University Hospital in Tübingen, Tübingen, Germany
- Sant Joan de Déu Barcelona Hospital, Esplugues de Llobregat, Barcelona, Spain
- National Taiwan University Hospital, Taipei, Taiwan
- Ankara University, Ankara, Turkey, Turkey (Türkiye)
- University College London, London, United Kingdom, United Kingdom